CLINICAL TRIAL: NCT04502225
Title: Impact of Decreased Venous Return on Supine Blood Pressure
Brief Title: Effect of Raised Head of the Bed on Lying Blood Pressure in Autonomic Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200124
Record Dates: First submitted 2020-07-20; First posted 2020-08-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Supine Hypertension; Autonomic Failure
MeSH Terms: conditions — Pure Autonomic Failure | interventions — Head-Down Tilt; Home Care Services

STUDY DESIGN:
Intervention Model Description: Randomized comparison of the effects of two amounts of head elevation (9 and 12 inches) achieved by tilting the bed or raising the head of the bed (up to four comparisons made) on supine blood pressure
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Elevation of the whole bed (tilt) (Experimental): Tilt of the whole bed so that the participant's head is raised by 9 and/or 12 inches.
  Interventions: Other: Tilt
- Elevation of the trunk (Experimental): Elevation of the trunk by tilting just the head of the bed so that the participant's head is raised by 9 and/or 12 inches.
  Interventions: Other: Elevated trunk
- Elevation of the whole bed (tilt) - In home (Experimental): Tilt of the whole bed so that the participant's head is raised by 8 inches.
  Interventions: Other: Tilt - In home
- Elevation of the trunk - In home (Experimental): Elevation of the trunk by raising the head 8 inches on a wedge pillow.
  Interventions: Other: Elevated Trunk - In home

INTERVENTIONS:
Other: Tilt — Tilt of the whole bed so that the head is elevated by 9 and/or 12 inches in an acute trial or overnight.
  Arms: Elevation of the whole bed (tilt)
Other: Elevated trunk — Elevation of the trunk through raising just the head of the bed until the head is elevated by 9 and/or 12 inches in an acute trial or overnight.
  Arms: Elevation of the trunk
Other: Tilt - In home — Tilt of the whole bed so that the head is elevated by 8 inches overnight.
  Arms: Elevation of the whole bed (tilt) - In home
Other: Elevated Trunk - In home — Elevation of the trunk through raising the head 8 inches on a wedge pillow overnight.
  Arms: Elevation of the trunk - In home

SUMMARY:
Many persons with autonomic failure often have high blood pressure when lying down (supine hypertension). This study is exploring the impact of decreased venous return to the heart (achieved by raising the head of the bed) to lessen supine blood pressure. If decreased venous return to the heart is effective at lowering supine blood pressure, these approaches may be utilized to treat supine hypertension non-pharmacologically. Raising the head of the bed decreases the amount of blood returning to the heart due to the effects of gravity. In this case, the decreased blood return to the heart may decrease blood pressure.

DETAILED DESCRIPTION:
Autonomic failure (AF) is a severely disabling condition, which is characterized by orthostatic hypotension (severe drop in blood pressure upon standing), bladder and bowel dysfunction, and sexual dysfunction. Besides disabling orthostatic hypotension, however, half of these patients have supine hypertension (high blood pressure when lying). Sustained high blood pressure is a cardiac risk for heart disease, kidney disease, and stroke. Sustained supine hypertension during the night induces pressure natriuresis (increased urine production due to high blood pressure) and volume loss (due to frequent urination/high volumes of urine), worsening orthostatic hypotension the following morning (blood pressure falls even more when the blood volume has been decreased due to loss of fluids in urine) and may also complicate the treatment of orthostatic hypotension with pressor agents (giving a blood pressure pill to prevent overnight high blood pressure may make daytime standing blood pressure worse).

Upright posture induces significant gravitational pooling of blood in the lower body that is normally compensated for by sympathetic activation. Failure of compensatory sympathetic activation results in orthostatic hypotension in autonomic failure patients due to the reduction in venous return and cardiac output. This abnormality has been used in autonomic failure patients with supine hypertension to their benefit by having them sleep with the head of the bed tilted up. The recommended amount of head up tilt is 10°, or about a 9-inch elevation of the head of the bed. In the investigators' hands this degree of tilt produces a significant but only modest decrease in blood pressure. Compliance is a limiting factor because most patients (and their spouses) are not able to tolerate even this modest level of head up tilt. Participants often elevate just the torso overnight, but the effect of this approach on supine blood pressure has not been reported.The investigators would like to compare the effects of tilt versus only elevating the head on supine blood pressure.

The existing knowledge provides the rationale for the study of the elevation of the head of the bed as a non-pharmacologic approaches for the treatment of supine hypertension in these patients. Elevation of the head of the bed will decrease venous return to the heart using the effects of gravity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with autonomic failure and with supine hypertension from all races
* Males and females, between 18 to 85 years

Exclusion Criteria:

* All medical students
* Pregnant women
* High-risk patients (for example: heart failure, symptomatic coronary artery disease, liver impairment, history of stroke or myocardial infarction)
* History of serious allergies or asthma.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-08-21 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 10 PM to 8 AM
  Maximal change from baseline in systolic blood pressure during the night
Systolic Blood Pressure | 10 PM to 8 AM or acute session (1 hour at each elevation of the head)
  Difference in systolic blood pressure between tilt and elevated trunk sessions

SECONDARY OUTCOMES:
Overnight Urine Volume | 10 PM to 8 AM
  Comparison of total urinary volume overnight.

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No